CLINICAL TRIAL: NCT01420627
Title: A Study of EZN-2279 (Polyethylene Glycol Recombinant Adenosine Deaminase [PEG-rADA]) Administered as a Weekly Intramuscular Injection in Patients With Adenosine Deaminase (ADA)-Deficient Combined Immunodeficiency
Brief Title: EZN-2279 in Patients With ADA-SCID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STP-2279-002
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: ADA-SCID; Adenosine Deaminase Deficiency; Severe Combined Immunodeficiency
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency; Severe Combined Immunodeficiency | interventions — pegademase bovine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adagen/EZN-2279 (Experimental): Patients started on Adagen and crossed over to experimental EZN-2279 treatment after at least a 3 week Lead-in Period on Adagen
  Interventions: Biological: EZN-2279; Biological: Adagen

INTERVENTIONS:
Biological: EZN-2279 — Weekly administration of EZN-2279 via IM injection
  Other Names: rADA
Biological: Adagen

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and pharmacokinetics of EZN-2279 in patients with ADA-deficient combined immunodeficiency currently being treated with Adagen.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ADA-deficient combined immunodeficiency
2. Stable clinical status while receiving therapy with Adagen®. Patients previously receiving gene therapy or undergoing hematopoietic stem cell transplantation who still require Adagen® treatment are eligible. The dose of Adagen® must be stable for at least 6 months prior to study entry.
3. Have both of the following during the Adagen® Lead-in phase of the study prior to EZN-2279 transition:

   1. Trough plasma ADA activity >15 μmol/h/mL while receiving Adagen® and
   2. Total erythrocyte dAXP ≤0.02 μmol/mL from a trough blood sample
4. Patients or parent/guardian must be capable of understanding the protocol requirements and risks and providing written informed assent/consent

Exclusion Criteria:

1. Autoimmunity requiring immunosuppressive treatment
2. Patients with detectable neutralizing anti-Adagen® antibodies at screening evaluation
3. Severe thrombocytopenia (platelet count <50 x 10^9/L)
4. Current participation in other therapeutic protocols for ADA-deficient combined immunodeficiency
5. Current or prior participation in another clinical study with an investigational agent and/or use of an investigational drug in the 30 days before study entry
6. Known planned participation in a gene-therapy study for the planned duration of this study
7. Any condition that, in the opinion of the PI, makes the patient unsuitable for the study
8. Inability or unwillingness to administer Adagen® or EZN-2279 on a one-time-per-week regimen
9. Inability to comply with the study protocol
10. Female patients who are pregnant or lactating
11. Female patients who are breast-feeding
12. Female subjects of childbearing potential who are not using an FDA approved birth control method

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elie Haddad, MD, PhD, Principal Investigator — Université de Montréal
Locations (6):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - UBMD, Buffalo, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Penn State College of Medicine The Milton S. Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adagen/EZN-2279: Patients started on Adagen and crossed over to experimental EZN-2279 treatment
Period: Adagen Lead-in Period
Arm/Group | Adagen/EZN-2279
Started (3 weeks, minimum) | 7
Completed | 7
Not Completed | 0
Period: EZN-2279 Treatment Period
Arm/Group | Adagen/EZN-2279
Started (Weeks T-1 through T-21) | 7
Completed | 6
Not Completed | 1
Not completed — Adverse Event | 1
Period: EZN-2279 Maintenance Period
Arm/Group | Adagen/EZN-2279
Started (Continuing until end of study, at least 203 weeks) | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: As-treated
Groups:
- Adagen/EZN-2279: Patients started on Adagen and crossed over to experimental EZN-2279 treatment after at least a 3 week Lead-in Period on Adagen
  EZN-2279: Weekly administration of EZN-2279 via IM injection
  Adagen
Arm/Group | Adagen/EZN-2279
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Detoxified At Each Visit in EZN-2279 Treatment Period
Description: Number of patients with total erythrocyte dAXP concentration from a trough blood sample <0.02 mmol/L
Time Frame: Baseline through Week T-21
Population: Completer
Measure: Count of Participants; unit: Participants
Groups:
- EZN-2279: Patients received EZN-2279 following at least a 3-week Lead-in Period with Adagen
Arm/Group | EZN-2279
Number analyzed (Participants) | 6
Participants
  Baseline | 6
  Week T-1 | 6
  Week T-3 | 6
  Week T-5: number analyzed (Participants) | 5
  Week T-5 | 5
  Week T-7 | 6
  Week T-8 | 6
  Week T-9: number analyzed (Participants) | 3
  Week T-9 | 3
  Week T-10: number analyzed (Participants) | 5
  Week T-10 | 5
  Week T-11 | 6
  Week T-13 | 6
  Week T-15 | 6
  Week T-17 | 6
  Week T-19 | 6
  Week T-21 | 6

2. Secondary Outcome: Safety Summary Data
Description: Summary of adverse events and serious adverse events
Time Frame: Through end of EZN-2279 study treatment, up to 203 weeks
Population: As-treated
Measure: Count of Participants; unit: Participants
Groups:
- Adagen: Patients received Adagen during the Lead-in Period
- EZN-2279: Patients received EZN-2279 after crossing over from at least a 3 week Adagen Lead-in
Arm/Group | Adagen | EZN-2279
Number analyzed (Participants) | 7 | 7
Participants
  Patients with treatment-emergent adverse events | 6 | 7
  Mild TEAE | 4 | 1
  Moderate TEAE | 2 | 3
  Severe TEAE | 0 | 3
  Treatment-related adverse event | 1 | 2
  Mild related AE | 1 | 1
  Moderate related AE | 0 | 0
  Severe related AE | 0 | 1
  Patients with any SAE | 0 | 4
  Patients discontinued treatment due to AE | 0 | 1
  Non-serious AEs | 6 | 7

3. Secondary Outcome: Summary of Trough ADA Activity Levels in EZN-2279 Treatment Period
Description: Trough ADA activity, mmol/h/L
Time Frame: From Baseline through Week T-21
Population: Completer
Measure: Median (Full Range); unit: mmol/h/L
Groups:
- EZN-2279 Treatment Period: Patients who completed at least a 3-week Adagen Lead-in Period and entered the 21-week Treatment Period
Arm/Group | EZN-2279 Treatment Period
Number analyzed (Participants) | 6
mmol/h/L
  Baseline | 15.7800 [13.200 to 22.900]
  Week T-1 | 14.0950 [9.130 to 24.600]
  Change from Baseline at Week T-1 | -1.7450 [-8.000 to 5.000]
  Week T-3 | 23.3850 [11.860 to 30.200]
  Change from Baseline at Week T-3 | 7.6500 [-4.060 to 9.360]
  Week T-5: number analyzed (Participants) | 5
  Week T-5 | 28.5600 [25.900 to 33.040]
  Change from Baseline at Week T-5: number analyzed (Participants) | 5
  Change from Baseline at Week T-5 | 13.3800 [3.000 to 17.400]
  Week T-7 | 34.8000 [29.240 to 42.590]
  Change from Baseline at Week T-7 | 19.000 [11.000 to 26.950]
  Week T-8 | 32.9300 [29.200 to 48.700]
  Change from Baseline at Week T-8 | 18.7400 [6.300 to 29.100]
  Week T-9: number analyzed (Participants) | 3
  Week T-9 | 38.8750 [26.160 to 52.800]
  Change from Baseline at Week T-9: number analyzed (Participants) | 3
  Change from Baseline at Week T-9 | 24.6840 [9.600 to 33.200]
  Week T-10: number analyzed (Participants) | 5
  Week T-10 | 37.7000 [23.480 to 46.200]
  Change from baseline at Week T-10: number analyzed (Participants) | 5
  Change from baseline at Week T-10 | 24.5000 [6.100 to 28.280]
  Week T-11 | 36.4350 [19.290 to 44.850]
  Change from Baseline at Week T-11 | 21.1950 [3.370 to 29.210]
  Week T-13 | 36.1000 [18.930 to 55.180]
  Change from Baseline at Week T-13 | 21.1150 [3.010 to 39.540]
  Week T-15 | 35.7850 [26.150 to 43.300]
  Change from Baseline at Week T-15 | 20.3950 [10.230 to 26.970]
  Week T-17 | 31.1000 [24.040 to 63.590]
  Change from Baseline at Week T-17 | 12.3500 [8.120 to 47.950]
  Week T-19 | 32.4200 [24.350 to 55.030]
  Change from Baseline at Week T-19 | 14.4300 [6.500 to 39.390]
  Week T-21 | 30.1500 [23.860 to 43.930]
  Change from Baseline at Week T-21 | 13.7500 [5.300 to 28.290]

4. Secondary Outcome: Summary of Trough ADA Activity Levels in EZN-2279 Maintenance Period
Description: Trough ADA activity levels, mmol/h/L
Time Frame: Through end of EZN-2279 study treatment, up to 203 weeks
Population: Completer
Measure: Median (Full Range); unit: mmol/h/L
Arm/Group | EZN-2279 Treatment Period
Number analyzed (Participants) | 6
mmol/h/L
  Baseline | 15.7800 [13.200 to 22.900]
  Week 34 | 31.1000 [16.400 to 51.800]
  Change from Baseline at Week 34 | 14.0350 [0.480 to 36.160]
  Week 47 | 37.9000 [16.170 to 42.230]
  Change from Baseline at Week 47 | 21.2600 [0.250 to 26.590]
  Week 60: number analyzed (Participants) | 3
  Week 60 | 35.3100 [13.440 to 50.770]
  Change from Baseline at Week 60: number analyzed (Participants) | 3
  Change from Baseline at Week 60 | 20.1300 [-2.480 to 35.130]
  Week 73: number analyzed (Participants) | 5
  Week 73 | 42.1900 [31.250 to 47.550]
  Change from Baseline at Week 73: number analyzed (Participants) | 5
  Change from Baseline at Week 73 | 22.5900 [15.330 to 34.350]
  Week 86: number analyzed (Participants) | 5
  Week 86 | 41.2000 [24.870 to 54.960]
  Change from Baseline at Week 86: number analyzed (Participants) | 5
  Change from Baseline at Week 86 | 25.5600 [8.950 to 41.760]
  Week 99: number analyzed (Participants) | 5
  Week 99 | 42.200 [27.330 to 57.090]
  Change from Baseline at Week 99: number analyzed (Participants) | 5
  Change from Baseline at Week 99 | 26.5800 [4.430 to 37.490]
  Week 112: number analyzed (Participants) | 4
  Week 112 | 31.6750 [23.340 to 44.840]
  Change from Baseline at Week 112: number analyzed (Participants) | 4
  Change from Baseline at Week 112 | 10.4250 [7.420 to 31.640]
  Week 125: number analyzed (Participants) | 4
  Week 125 | 39.2700 [33.300 to 44.990]
  Change from Baseline at Week 125: number analyzed (Participants) | 4
  Change from Baseline at Week 125 | 21.1150 [11.190 to 31.790]
  Week 138: number analyzed (Participants) | 3
  Week 138 | 46.0600 [31.850 to 51.820]
  Change from Baseline at Week 138: number analyzed (Participants) | 3
  Change from Baseline at Week 138 | 26.4600 [8.950 to 38.620]
  Week 151: number analyzed (Participants) | 3
  Week 151 | 36.6700 [30.370 to 44.890]
  Change from Baseline at Week 151: number analyzed (Participants) | 3
  Change from Baseline at Week 151 | 17.070 [7.470 to 31.690]
  Week 164: number analyzed (Participants) | 3
  Week 164 | 34.4500 [27.950 to 41.990]
  Change from Baseline at Week 164: number analyzed (Participants) | 3
  Change from Baseline at Week 164 | 11.5500 [8.350 to 28.790]
  Week 177: number analyzed (Participants) | 3
  Week 177 | 33.1300 [26.980 to 47.850]
  Change from Baseline at Week 177: number analyzed (Participants) | 3
  Change from Baseline at Week 177 | 13.5300 [4.080 to 34.650]
  Week 190: number analyzed (Participants) | 3
  Week 190 | 32.5000 [31.180 to 38.920]
  Change from Baseline at Week 190: number analyzed (Participants) | 3
  Change from Baseline at Week 190 | 11.5800 [9.600 to 25.720]
  Week 203: number analyzed (Participants) | 3
  Week 203 | 36.3300 [33.890 to 43.310]
  Change from Baseline at Week 203: number analyzed (Participants) | 3
  Change from Baseline at Week 203 | 16.7300 [10.990 to 30.110]
  End of Study/Early Discontinuation: number analyzed (Participants) | 3
  End of Study/Early Discontinuation | 39.7700 [33.740 to 46.170]
  Change from Baseline at End of Study/Early Discont: number analyzed (Participants) | 3
  Change from Baseline at End of Study/Early Discont | 22.3800 [10.840 to 30.530]

5. Secondary Outcome: Summary of Trough dAXP Levels in EZN-2279 Treatment Period
Description: Trough dAXP levels, mmol/L
Time Frame: From Baseline through Week T-21
Population: Completer
Measure: Median (Full Range); unit: mmol/L
Arm/Group | EZN-2279 Treatment Period
Number analyzed (Participants) | 6
mmol/L
  Baseline | 0.0020 [0.002 to 0.002]
  Week T-1 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-1 | 0.0000 [0.000 to 0.000]
  Week T-3 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-3 | 0.0000 [0.000 to 0.000]
  Week T-5: number analyzed (Participants) | 5
  Week T-5 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-5: number analyzed (Participants) | 5
  Change from Baseline at Week T-5 | 0.0000 [0.000 to 0.000]
  Week T-7 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-7 | 0.0000 [0.000 to 0.000]
  Week T-8 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-8 | 0.0000 [0.000 to 0.000]
  Week T-9: number analyzed (Participants) | 3
  Week T-9 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-9: number analyzed (Participants) | 3
  Change from Baseline at Week T-9 | 0.0000 [0.000 to 0.000]
  Week T-10: number analyzed (Participants) | 5
  Week T-10 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-10: number analyzed (Participants) | 5
  Change from Baseline at Week T-10 | 0.0000 [0.000 to 0.000]
  Week T-11 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-11 | 0.0000 [0.000 to 0.000]
  Week T-13 | 0.0020 [0.002 to 0.032]
  Change from Baseline at Week T-13 | 0.0000 [0.000 to 0.030]
  Week T-15 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-15 | 0.0000 [0.000 to 0.000]
  Week T-17 | 0.0020 [0.002 to 0.047]
  Change from Baseline at Week T-17 | 0.0000 [0.000 to 0.045]
  Week T-19 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-19 | 0.0000 [0.000 to 0.000]
  Week T-21 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week T-21 | 0.0000 [0.000 to 0.000]

6. Secondary Outcome: Summary of Trough dAXP Levels in EZN-2279 Maintenance Period
Description: Trough dAXP levels, mmol/L
Time Frame: Through end of EZN-2279 study treatment, up to 203 weeks
Population: Completer
Measure: Median (Full Range); unit: mmol/L
Arm/Group | EZN-2279 Treatment Period
Number analyzed (Participants) | 6
mmol/L
  Baseline | 0.0020 [0.002 to 0.002]
  Week 34 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week 34 | 0.0000 [0.000 to 0.000]
  Week 47 | 0.0020 [0.002 to 0.008]
  Change from Baseline at Week 47 | 0.0000 [0.000 to 0.006]
  Week 60: number analyzed (Participants) | 3
  Week 60 | 0.0020 [0.002 to 0.008]
  Change from Baseline at Week 60: number analyzed (Participants) | 3
  Change from Baseline at Week 60 | 0.0000 [0.000 to 0.006]
  Week 73: number analyzed (Participants) | 5
  Week 73 | 0.0020 [0.002 to 0.006]
  Change from Baseline at Week 73: number analyzed (Participants) | 5
  Change from Baseline at Week 73 | 0.0000 [0.000 to 0.004]
  Week 86: number analyzed (Participants) | 5
  Week 86 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week 86: number analyzed (Participants) | 5
  Change from Baseline at Week 86 | 0.0000 [0.000 to 0.000]
  Week 99: number analyzed (Participants) | 5
  Week 99 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week 99: number analyzed (Participants) | 5
  Change from Baseline at Week 99 | 0.000 [0.000 to 0.000]
  Week 112: number analyzed (Participants) | 4
  Week 112 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week 112: number analyzed (Participants) | 4
  Change from Baseline at Week 112 | 0.0000 [0.000 to 0.000]
  Week 125: number analyzed (Participants) | 4
  Week 125 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week 125: number analyzed (Participants) | 4
  Change from Baseline at Week 125 | 0.0000 [0.000 to 0.000]
  Week 138: number analyzed (Participants) | 3
  Week 138 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week 138: number analyzed (Participants) | 3
  Change from Baseline at Week 138 | 0.0000 [0.000 to 0.000]
  Week 151: number analyzed (Participants) | 3
  Week 151 | 0.0020 [0.002 to 0.005]
  Change from Baseline at Week 151: number analyzed (Participants) | 3
  Change from Baseline at Week 151 | 0.0000 [0.000 to 0.003]
  Week 164: number analyzed (Participants) | 3
  Week 164 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week 164: number analyzed (Participants) | 3
  Change from Baseline at Week 164 | 0.0000 [0.000 to 0.000]
  Week 177: number analyzed (Participants) | 3
  Week 177 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week 177: number analyzed (Participants) | 3
  Change from Baseline at Week 177 | 0.0000 [0.000 to 0.000]
  Week 190: number analyzed (Participants) | 3
  Week 190 | 0.0020 [0.002 to 0.002]
  Change from Baseline at Week 190: number analyzed (Participants) | 3
  Change from Baseline at Week 190 | 0.0000 [0.000 to 0.000]
  Week 203: number analyzed (Participants) | 3
  Week 203 | 0.0020 [0.002 to 0.008]
  Change from Baseline at Week 203: number analyzed (Participants) | 3
  Change from Baseline at Week 203 | 0.0000 [0.000 to 0.006]
  End of Study/Early Discontinuation | 0.0020 [0.002 to 0.010]
  Change from Baseline at End of Study/Early Discont | 0.0000 [0.000 to 0.008]

7. Secondary Outcome: Number of Patients With Infections and Hospitalizations
Description: Infections were documented clinically with signs and symptoms without microbiologic cultures or with positive viral or bacterial cultures
Time Frame: Through end of EZN-2279 study treatment, up to 203 weeks
Population: As-treated
Measure: Count of Participants; unit: Participants
Arm/Group | EZN-2279
Number analyzed (Participants) | 7
Participants
  Patients with infection | 5
  Patients with hospitalizations | 3

8. Secondary Outcome: Duration of Hospitalization
Time Frame: Through end of EZN-2279 study treatment, up to 203 weeks
Population: As-treated population who were hospitalized
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Number of hospitalizations (3 patients)
Arm/Group | EZN-2279
Number analyzed (Participants) | 3
Number analyzed (Number of hospitalizations (3 patients)) | 4
Days | 5.0 (2.16)

9. Secondary Outcome: Number of Patients Detoxified At Each Visit in EZN-2279 Maintenance Period
Description: Number of patients with total erythrocyte dAXP concentration from a trough blood sample <0.02 mmol/L
Time Frame: From Week 34 to End of Study/Early Discontinuation, up to 203 weeks
Population: Completer
Measure: Count of Participants; unit: Participants
Arm/Group | EZN-2279 Treatment Period
Number analyzed (Participants) | 6
Participants
  Baseline | 6
  Week 34 | 6
  Week 47 | 6
  Week 60 | 3
  Week 73: number analyzed (Participants) | 5
  Week 73 | 5
  Week 86: number analyzed (Participants) | 5
  Week 86 | 5
  Week 99: number analyzed (Participants) | 5
  Week 99 | 5
  Week 112: number analyzed (Participants) | 4
  Week 112 | 4
  Week 125: number analyzed (Participants) | 4
  Week 125 | 4
  Week 138: number analyzed (Participants) | 3
  Week 138 | 3
  Week 151: number analyzed (Participants) | 3
  Week 151 | 3
  Week 164: number analyzed (Participants) | 3
  Week 164 | 3
  Week 177: number analyzed (Participants) | 3
  Week 177 | 3
  Week 190: number analyzed (Participants) | 3
  Week 190 | 3
  Week 203: number analyzed (Participants) | 3
  Week 203 | 3
  End of Study/Early Discontinuation: number analyzed (Participants) | 3
  End of Study/Early Discontinuation | 3

ADVERSE EVENTS:
Time Frame: Through end of EZN-2279 study treatment, up to 203 weeks
Groups:
- Adagen: Patients received Adagen during the Lead-in Period (at least 3 weeks)
- EZN-2279: Patients received EZN-2279 after crossing over from Adagen
Arm/Group | Adagen | EZN-2279
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 4/7
Other Adverse Events (participants affected / at risk) | 6/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adagen (N=7) | EZN-2279 (N=7)
Respiratory tract infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Vestibular migraine (Nervous system disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adagen (N=7) | EZN-2279 (N=7)
Non-cardiac chest pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Injection site bruising (General disorders) | 0 | 1
Injection site discomfort (General disorders) | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Nodule (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Alveolar osteitis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 1
Ear lobe infection (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Genital infection fungal (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 1
Haemophilus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Stoma site infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Epidermodysplasia verruciformis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Vestibular migraine (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Blood immunoglobulin G increased (Investigations) | 0 | 1
Immunoglobulins increased (Investigations) | 0 | 1
Monoclonal immunoglobulin present (Investigations) | 0 | 1
Crystal urine present (Investigations) | 1 | 0
Full blood count abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Scrotal mass (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Superior vena cava stenosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT01420627/SAP_000.pdf
  • Study Protocol (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT01420627/Prot_001.pdf